CLINICAL TRIAL: NCT02438943
Title: A Cluster Randomized Controlled Trial of an Intervention to Improve the Management of Dyslipidemia in Primary Care
Brief Title: An Intervention to Improve Management of Dyslipidemia in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ECP218,11/12
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Cardiovascular Disease; Dyslipidemia; Diabetes Melletus; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Audit and Physician intervention (Active Comparator): The intervention will comprise the feedback of the results of the baseline audit, training in motivational interviewing for clinic staff, use of a physician reminder stamp in the patients' charts and distribution of patient education cards
  Interventions: Other: Audit; Other: Physician Intervention
- Audit only (Sham Comparator): The intervention will comprise the feedback of the results of the baseline audit only
  Interventions: Other: Audit

INTERVENTIONS:
Other: Audit — An assessment of medical records using a pre-specified audit instrument to assess the level of care given for clinic attendees with cardiovascular disease including dyslipidemia
Other: Physician Intervention — Feedback Training sessions for physicians inclusive Motivational Interviewing training and the use of physician reminders on medical records before each clinic session
  Arms: Audit and Physician intervention

SUMMARY:
To assess the effectiveness of a clinical audit and physician based intervention in improving the management of dyslipidemia at Health centres in the Southeast Health Region of Jamaica

ELIGIBILITY:
Inclusion Criteria:

* Attended the clinic for at least 18 months
* Is diagnosed with any of hypertension, diabetes, dyslipidemia, stroke, coronary heart disease (including angina, myocardial infarction), congestive cardiac failure or peripheral arterial disease, were eligible to be included in the audit

Exclusion Criteria:

* acutely ill or was diagnosed with established kidney disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of persons attending health centers in the Southeast Health region with normal lipid values | 1 year

SECONDARY OUTCOMES:
Proportion of persons attending health centers in the Southeast Health region with normal glucose values | 1 year
Proportion of persons attending health centers in the Southeast Health region with normal blood pressure values | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of the West Indies, mona, Kingston, Jamaica